CLINICAL TRIAL: NCT04697797
Title: Mechanical and Electrical Dyssynchrony During His-Bundle Pacing (Selective and Non-selective) Versus His-Bundle Area Right Ventricular Pacing
Brief Title: Mechanical and Electrical Dyssynchrony During His-Bundle Pacing Versus His-Bundle Area Right Ventricular Pacing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Other Study IDs: RNN/147/20/KE
Record Dates: First submitted 2020-12-14; First posted 2021-01-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Bradyarrhythmia
Keywords: His Bundle Pacing; Dyssynchrony; Echocardiography; ECG
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Device Programming — Intervention includes (1) pacemaker reprogramming (2) echocardiographic parameters acquisition (3) ECG recording
  Other Names: Echocardiography; ECG

SUMMARY:
The aim of this study is to evaluate mechanical and electrical cardiac dyssynchrony in patients with pacemakers and the right ventricular electrode implanted in His Bundle area.

DETAILED DESCRIPTION:
Permanent His Bundle Pacing (HBP) is a well-known method of cardiac pacing which is increasingly used in everyday practice. After lead implantation in His Bundle area (HBA) capture of various tissues can be achieved: A. right ventricular myocardium near to HBP; B. cardiac conduction system selectively or nonselectively (with concomitant regional myocardium activation). The different excitability and refractory periods decide which tissue, myocardium or/and the conduction system is effectively paced. A lot of clinical trials revealed the advantage of HBP over apical ventricular pacing (AVP). HBP improves clinical (NYHA, quality of life, hospitalization rate) and echocardiographic (left ventricular dimension and ejection fraction) indicators of heart failure.

We are going to compare mechanical and electrical synchrony during the various type of myocardium activation: HBP (nsHBP or sHBP), RV pacing near HBA and native heart rhythm (if possible) in each patient recruited to the study. Adequate pacemaker programming will allow achieving different activations as shown above. The mechanical synchrony will be estimated by transthoracic echocardiography and the electrical one by the detailed analysis of ECG.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients after implantation of pacemaker system with pacing lead successfully captured His Bundle (selectively or/and nonselectively)

Exclusion Criteria:

* not willing or incapable to give written informed consent;
* previous implanted cardiac electronic device (pacemaker, implantable cardioverter-defibrillator, cardiac resynchronization therapy device)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bradyarrhythmia and indications for de novo permanent pacemaker implantation. The decision for pacing lead placement in His Bundle is left for physician discretion. Patients after pacemaker system implantation with His Bundle successfully pacing are to be asked to participate in the study. After having written informed consent obtained patients are to be scheduled for ventricular synchrony evaluation with ECHO and ECG after 3-6 months after implant (mid-term) and after 12 months (long-term).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Interventricular mechanical delay | Mid-term: 3-6 months after pacemaker implantation
  InterVentricular Mechanical Dyssynchrony Parameter 1
Interventricular mechanical delay | Long term: 12-15 months after pacemaker implantation
  InterVentricular Mechanical Dyssynchrony Parameter 1
Free-wall-LV-to-RV-delay | Mid-term: 3-6 months after pacemaker implantation
  InterVentricular Mechanical Dyssynchrony Parameter 2
Free-wall-LV-to-RV-delay | Long term: 12-15 months after pacemaker implantation
  InterVentricular Mechanical Dyssynchrony Parameter 2
Septal-to-posterior wall motion delay | Mid-term: 3-6 months after pacemaker implantation
  IntraVentricular Mechanical Dyssynchrony Parameter 1
Septal-to-posterior wall motion delay | Long term: 12-15 months after pacemaker implantation
  IntraVentricular Mechanical Dyssynchrony Parameter 1
Opposing wall motion delay | Long term: 12-15 months after pacemaker implantation
  IntraVentricular Mechanical Dyssynchrony Parameter 2
Opposing wall motion delay | Mid-term: 3-6 months after pacemaker implantation
  IntraVentricular Mechanical Dyssynchrony Parameter 2
systolic dyssynchrony index | Long term: 12-15 months after pacemaker implantation
  Ventricular Mechanical Dyssynchrony Parameter 1
systolic dyssynchrony index | Mid-term: 3-6 months after pacemaker implantation
  Ventricular Mechanical Dyssynchrony Parameter 1
QRS duration | Mid-term: 3-6 months after pacemaker implantation
  Electrical dyssynchrony Parameter
QRS duration | Long term: 12-15 months after pacemaker implantation
  Electrical dyssynchrony Parameter

SECONDARY OUTCOMES:
Radial strain | Mid-term: 3-6 months after pacemaker implantation
  Additional Ventricular Mechanical Dyssynchrony Parameter 1
Radial strain | Long term: 12-15 months after pacemaker implantation
  Additional Ventricular Mechanical Dyssynchrony Parameter 1
Left Ventricular Ejection Fraction | Mid-term: 3-6 months after pacemaker implantation
  Global left ventricle function parameter
Left Ventricular Ejection Fraction | Long term: 12-15 months after pacemaker implantation
  Global left ventricle function parameter
Global longitudinal strain | Mid-term: 3-6 months after pacemaker implantation
  Global left ventricle function parameter 2
Global longitudinal strain | Long term: 12-15 months after pacemaker implantation
  Global left ventricle function parameter 2
Left ventricular output track velocity-time integral | Mid-term: 3-6 months after pacemaker implantation
  Global left ventricle function parameter 3
Left ventricular output track velocity-time integral | Long term: 12-15 months after pacemaker implantation
  Global left ventricle function parameter 3
Diastolic Filling Time | Mid-term: 3-6 months after pacemaker implantation
  Atrioventricular Dyssynchrony Parameter
Diastolic Filling Time | Long term: 12-15 months after pacemaker implantation
  Atrioventricular Dyssynchrony Parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Electrocardiology Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided